CLINICAL TRIAL: NCT06477393
Title: The Inclusion of Natural Healing Factors in Complex Regular Rehabilitation of Patients with Degenerative Small Joints Disease: Impact on Changes in Functional Status, Quality of Life, and Socio-economic Significance in Reducing Temporary Incapacity for Work and Disability, Improving Participation
Brief Title: Balneotherapy and Peloid Therapy Impact Small Joint Diseases
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Versmė (Unknown)
Responsible Party: Principal Investigator, Ona Montvydaite-Kreivaitiene, PhD Candidate, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V-2
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis; Hand Osteoarthritis; Foot Osteoarthritis
Keywords: balneotherapy, peloid therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Baths; Balneology

STUDY DESIGN:
Intervention Model Description: The study employs a parallel-group design, where participants are randomly assigned to one of two groups: an experimental group receiving the enhanced rehabilitation program with natural healing factors and a control group receiving the standard rehabilitation program. The randomisation ensures that each participant has an equal chance of being assigned to either group, minimising selection bias and ensuring comparability between the groups.
Who Masked: Investigator
Masking Description: The participants can guess indirectly, and the main researcher, the laboratory investigator, will be blind to the group assignments. This single-blinded design is chosen to facilitate the implementation and adherence to the rehabilitation programs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): The control group will receive "placebo" type procedures in addition to the usual medical rehabilitation procedures, i.e., heat treatments, so routine health care will not be lost. The typical procedures are assigned in accordance with the order of the Minister of Health of the Republic of Lithuania "On the approval of descriptions of general and special requirements for the provision of medical rehabilitation and anti-recidivism sanatorium treatment services" valid version dated 06.14.2023). In-resort sanatoriums, the mud and mineral water procedures are additionally paid services, which the sanatorium will provide free of charge for scientific development.
  Interventions: Other: Regular rehababilitation; Other: Heat procedures
- Experimental group (Active Comparator): Standard rehabilitation procedures will be applied (following the order of the Minister of Health of the Republic of Lithuania) supplemented by balneotherapy/peloid therapy. Rehabilitation procedures will be performed in the Lithuanian resort Birstonas sanatorium "Versme." The standard rehabilitation procedures will be the same as those in the control group.
  Interventions: Other: Regular rehababilitation; Other: Healing mud application; Other: Mineral water bath

INTERVENTIONS:
Other: Regular rehababilitation — Subjects of the experimental and control groups will receive routine procedures applied in the resort sanatorium: physiotherapy (28-32), occupational therapy (12-18), dry hydromassage (7-8), psychotherapy or audiovisual relaxation (3-4), social worker's visit ( 1-2), physiotherapy (magnetotherapy, ultrasound therapy (8-9).
  Other Names: Standart pysiotherapy
Other: Heat procedures — The bath is filled with 200 litres of warm tap water at 36-38°C. The participant lies in the prepared bath, ensuring the chest area remains uncovered. While in the bath, the participant performs gentle movements. The procedure lasts 12-15 minutes. Air is pumped into the water to increase the oxygen saturation in the bath environment.
  A prepared gel pack will be placed in another bag and heated to 50-55°C. The heated pack will be delivered to the treatment area using pumps. For applications, the gel pack is used at 40-42°C. Temperature of the gel pack can range between 38-43°C.
  Other Names: Bathing in tap water, hot packs
  Arms: Control group
Other: Healing mud application — Therapeutic mud applications: peat brought from the quarry is sifted, ground, and mixed with natural mineralisation of 20-22g/l with mineral water in a ratio of at least 4:1 until the consistency of thick sour cream. The prepared peat mud is heated to 50-55 degrees. The heated mud is fed to the place where the procedures are performed with the help of pumps. Mud mass at 40-42 degrees is used for applications. A mud temperature range of 38-43 degrees is possible.
  Before the procedure, it is recommended not to eat, go to the toilet, or take a warm shower. A polyethene film is laid on a special heated couch, and a 2-4 cm thick layer of mud is poured into the area of the hands and feet, covered with a blanket. After the procedure, the subject takes a warm, lukewarm shower, wipes himself with a soft towel, and rests. Peloids are not reused.
  Other Names: Peloid thearapy
  Arms: Experimental group
Other: Mineral water bath — The pearl bath is prepared by a physical method. The bath is filled with 200 l of warm 36-38 C mineral water, the subject lies in the prepared bath, leaving the heart area open, while lying in the bath he performs light movements. The duration of the procedure is 12-15 minutes. Air is blown into the water, which increases oxygen saturation in the bath environment. Before the procedure, it is recommended not to eat, go to the toilet, take a warm shower. After the procedure, the subject takes a warm, lukewarm shower, wipes himself with a soft towel and rests. Mineral waters are not reused.
  Other Names: Balneotherapy
  Arms: Experimental group

SUMMARY:
This clinical trial investigates the effects of natural healing factors (mineral water and mud procedures) in combination with regular rehabilitation of patients with degenerative small joint disease. The study aims to assess the impact on functional status, quality of life, and socio-economic factors, including the reduction of temporary incapacity for work and disability and the improvement of patient participation. Participants will undergo a regular rehabilitation program incorporating these natural healing factors, measuring outcomes through various health metrics.

DETAILED DESCRIPTION:
This interventional clinical trial is designed to evaluate the efficacy of incorporating natural healing factors into the standard rehabilitation regimen for patients suffering from degenerative small joint disease. The study will involve a well-defined cohort of participants diagnosed with this condition, randomly assigned to either the experimental group, which will receive the combination of mineral water and mud procedures with a regular rehabilitation program, or the control group, which will receive the standard regular rehabilitation.

The primary objective is to determine patients' functional status and quality of life changes, measured through validated health questionnaires and functional tests specific to small joints. Secondary objectives include analysing the socio-economic impact, reducing temporary incapacity for work and disability rates and improving patient participation in daily activities and employment.

The data collection process will be rigorous, involving a comprehensive mix of qualitative and quantitative methods. Participants will be required to complete health surveys and functional status tests and provide socioeconomic data at multiple points throughout the study. The rehabilitation program will include physiotherapy, occupational therapy, and the application of natural healing factors such as balneotherapy and peloid therapy.

ELIGIBILITY:
1. Inclusion Criteria:1. Adult (> 18 years).
2. Subjects will be diagnosed with symptomatic (duration greater than 3 months) osteoarthritis of the hands and/or feet and meet the validated classification or diagnostic criteria for hand and/or foot OA published by EULAR/ACR (Altman et al., 1990; Zhang et al. et al., 2009). Hand and/or foot joint pain at baseline will be at least 40 mm on a 100 mm visual analogue scale (VAS) (0 = no pain; 10 = worst pain) without pain medication.
3. Participants will be assessed for radiographic changes characteristic of osteoarthritis. This assessment will be based on the Kellgren-Lawrence (K-L) grading system, which is a widely used method for classifying the severity of osteoarthritis. The system is based on stages, with a minimum requirement of osteoarthritis in more than one joint and at least two stages of severity (Kellgren JH, 1957).
4. Rehabilitation procedures, except physical exercises performed at home, will not be applied for at least 2 months.
5. Subjects can sign the patient's informed consent form.

Exclusion Criteria:

1. Subjects with autoimmune diseases that can affect the joints of the hands/feet (rheumatoid arthritis, systemic connective tissue diseases, seronegative spondyloarthropathies) or crystalline arthropathies.
2. Diagnosed with thoracic outlet syndrome, carpal tunnel syndrome, Guyon's canal syndrome, cubital tunnel syndrome, diabetic neuropathy or cheiroarthropathy, palmar tenosynovitis, fibromyalgia and pain syndrome.
3. Subjects who have suffered serious injuries in the last 6 months or who have undergone surgical interventions on the joints of the hands/feet.
4. The functional tests provided in the study cannot be performed due to advanced OA or other diseases.
5. Subjects with skin lesions or sensitivity to the intended procedures.
6. Diagnosed with oncological diseases or being investigated for oncological diseases.
7. Diseases or conditions for which mud or mineral water baths are contraindicated
8. Constantly taking pain relievers for other conditions unless the dose is stable for ≥ 1 month.
9. Taking Sy-SADOA symptomatic slow-acting OA drugs unless the dose is stable for ≥ 3 months.
10. Pregnancy or planned pregnancy.
11. Intra-articular (IA) injection of corticosteroids (joints of hands and feet) within the last 1 month or IA injection of hyaluronic acid within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Heel-Rise Test | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  The Heel-Rise Test is a functional assessment used to evaluate the strength and endurance of the calf muscles, particularly the gastrocnemius and soleus muscles. During the test, the participant is asked to perform repeated heel rises while standing on one foot until they can no longer continue or until they reach a predetermined maximum number of repetitions. This test provides valuable information on muscle performance, which is critical for patients with degenerative small joints disease affecting the lower extremities. The outcome is measured by the number of heel rises completed and the quality of movement, including balance and control.
Pinch grip strength | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  The manometer will measure the finger compression force. This device will assess: first-second (I-II) finger grip strength, first-second-third (I-II-III) finger grip strength and grip strength. Evaluation units - kilograms (kg) Between muscle contraction measurements, a 30 s rest was applied in the bus to avoid the influence of muscle fatigue. The subjects will be evaluated with a manometer at each visit. Duration 3-5 min.
Hand grip strength | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  Hand grip muscle strength will be measured with a dynamometer. The dynamometer is held in the elbow-bent arm, away from the body. When evaluating with a dynamometer, the subject is seated, the shoulders are in a neutral position, the elbow is bent at an angle of 90°, the forearms are placed on the table, and the elbow deviation of the wrist is 0-15°. The device is pressed with maximum force, performing a single-hand pressing movement. The device is pressed with one hand and then with the other hand. The average of three clicks with the left and right hands is evaluated. The units of assessment are kilograms (kg). A 30 s rest will be applied between muscle contraction measurements to avoid the influence of muscle fatigue. A dynamometer will be used to assess subjects at each visit. Duration 5 min.
Hand Mobility in Scleroderma, HAMIS | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  Hand Mobility Test in Scleroderma (HAMIS) to assess osteoarthritis. The continuum consists of nine tasks that assess finger, thumb, and wrist mobility, with each task rated from 0 (no impairment) to 3 (cannot perform), resulting in a total possible score of 27 per hand. Standardised cylinders will assess finger flexion, finger extension and thumb adduction. The total score will be calculated as the average of the two hands (range 0-27). Finger and thumb mobility component scores will be calculated by summing the respective subscores: finger flexion, extension and abduction (range 0-9) for finger mobility, thumb adduction and pincer grasp (0-6) for thumb mobility. Duration 5-7 min.
Finger-to-palm, FTP | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  The finger-to-palm distance (FTP) will be measured. This measurement is important in assessing the mobility of the fingers and the possible limitation of movement due to various medical conditions such as osteoarthritis. Finger extension and flexion (maximal finger flexion and extension in all three finger joints: MKF, PIF and DIF) are measured.
Modified Kapandji Index, MKI | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  Based on anatomical landmarks, a Modified Kapandji (MKI) evaluation index will be performed, especially thumb opposition and finger flexion and extension movements. It allows you to assess the mobility of the fingers and thumb, giving a total score from 0 to 50, where lower scores indicate greater limitation of movement in one hand. The total score is obtained by summing the scores of the three items. Anatomical landmarks and scores are listed in Protocol Appendix No. 1. The total score will be calculated as the average of the two arms (range 0-50). Finger and thumb mobility components will be scored using the corresponding subscores: 2-5 finger flexion and extension (range 0-40) for finger mobility and thumb apposition (range 0-10) for thumb mobility. Duration 2-3 min. The test is performed at each visit.
Strength of extensor and flexor muscles of the foot | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  Strength of extensor and flexor muscles of the foot. The test uses a hand-held dynamometer. Strength is measured in kilograms. Force will be measured three times for each side, and the results will be averaged
ROM | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  The goniometer will measure the amplitudes during active movement: foot plantarflexion (bending), foot dorsiflexion (extension), and MTF dorsiflexion. The measurements will be repeated three times. The arithmetic mean is calculated after adding up all the results obtained during one measurement. The duration of the study is 5 minutes
30-second chair stand test | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  The maximum number of chair stand repetitions possible in a 30 second period
Stair climb test | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  The time (in seconds) it takes to ascend and descend a flight of stairs
40m (4x10m) fast-paced walk test | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft)
The single leg stance test SLS | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  This exercise is performed with eyes open and hands on hips. The subject stands on one leg without assistance; time starts when the opposite foot leaves the ground. Time stops immediately when the opposite foot touches the ground and/or when the hands leave the hips. It is repeated three times with both legs, and the average is evaluated. The duration is three minutes.
VAS | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months. Additionally, the VAS will be assessed for pain and stiffness each day before the procedures at 8-9 am. morning
  Patients' pain and stiffness will be assessed using a visual analogue (VAS) scale. Pain on squeezing MTF and MCF joints. VAS every day before procedures.
biomarkers | Before and after rehabilitation program
  Cytokines (IL-6, IL-1beta, and TNF alpha) and biochemical markers of cartilage (thrombospondin-5/COMP (Human Thrombospondin-5/COMP), aggrecan (PG)) will be performed using a standardised ELISA (English enzyme-linked immunosorbent assay) methodology.

SECONDARY OUTCOMES:
Manchester-Oxford Foot Questionnaire (MOxFQ) | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  MOxFQ measures foot pain, foot function and general foot health. The MOXFQ has three domains related to foot health: walking/standing problems (seven items), pain (five items), and problems with social relationships (four items). Duration: 5-10 minutes. The questionnaire has a Lithuanian version. Permission/license obtained for use.
Foot and ankle outcome score, FAOS | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  FAOS was designed to assess the patient's perception of their foot or ankle condition. The questionnaire consists of 5 subscales: pain, other symptoms, performance of daily activities tasks, function in sports and recreation, and ankle/foot-related quality of life questions. The subject answers the questions by describing the last week. Permission/license was obtained to prepare and use the Lithuanian version.
The Quality of life questionnaire SF-36 | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  SF-36 will be evaluated, which consists of 36 questions reflecting eight domains of life: physical activity, activity limitation due to physical ailments and emotional disturbances, social connections, emotional state, vigour/vitality, pain, and general health assessment. Each part is scored from 0 to 100 using a calculation algorithm. The higher the number, the better the quality of life. The questionnaire will be assessed at each visit. Duration: 10-15 minutes. The questionnaire was validated in Lithuanian in 2005. Cronbach alpha of Rugienė and co-authors=0.79-0.85. Permission received
The functional index for hand osteoarthritis FIHOA | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  FIHOA is a questionnaire designed to self-assess hand function in daily activities. Consists of 10 parts related to the function of the hands in daily activities. Each item is rated with four points on the Linkert scale. The subject rates his level of function from 0 (difficult) to 3 (impossible). Scores for each domain are cumulative: a higher score indicates more difficulty in performing daily activities. A total score of 0 indicates good performance, and 30 indicates poor hand activity. Duration about 3 minutes. Assessed at each visit. The author translated the questionnaire into Lithuanian. Freely available, no permission required, authors notified of study. Access: http://fihoa.net.
Michigan Hand Outcomes Questionnaire MHQ | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  The Michigan Questionnaire will assess the subject's independence and hand function. This questionnaire consists of 6 scales: general hand function, activity in daily activities, pain, work performance, aesthetic image of the hand, and opinion of the subject about his hand function. The subject evaluates the performance of each activity with points: the lowest (worst function) - 1 point, the highest (ideal function) - 5 points. The questionnaire consists of 72 questions. The authors' written consent was obtained. The questionnaire will be translated according to the standard methodology, and Cronbach's alpha coefficient will be checked.
Ultrasound of hand joints | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  Ultrasound examination of the hand joints will be performed based on the EULAR/OMERACT recommendations and according to Mario Giulini's protocol (D'Agostino et al., 2017; Giulini et al., 2023; Hammer et al., 2016). Ultrasound images of 26 joints of both hands will be evaluated. Synovitis, fluid, and osteophytes will be assessed. An ultrasound examination will be performed at each visit. Ultrasound images with initials are saved on the media.
Ultrasound of foot joints | Before the start of the rehabilitation program, follow up 2, 3, 6,12 months
  Ultrasound examination of the foot joints will be performed based on EULAR/OMERACT recommendations (G. A. Bruyn et al., 2019; G. A. W. Bruyn et al., 2019; Zabotti et al., 2019). Ultrasound examination will be an assessment in standard positions. 7 joints of both feet will be evaluated. Synovitis, fluid, and osteophytes will be assessed. An ultrasound examination will be performed at each visit. Ultrasound images with initials are saved on the media.

OTHER OUTCOMES:
Investigator's questionnaire | Before procedures
  The researcher will prepare a questionnaire on socio-demographic and anamnestic data, which will be evaluated (e.g., the degree of osteoarthritis, use of other drugs, co-morbidities, trauma and/or surgery in the past, use of physical factors in the hands and feet in the past.
x ray of joints | Before procedures
  Radiographs of the hands and feet will be evaluated (the test will already be performed on the subjects before they are included in the biomedical study). X-rays - images with initials and numbers are recorded on the medium.
BMI | Before procedures
  height and weight will be measured and body mass index will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Raimondas Kubilius, Prof, Principal Investigator — The Hospital of Lithuanian University of Health Sciences (LSMU) Kaunas clinics
Locations (2):
- Lithuania (2):
  - AB Birštonas health resort "Versmė", Birštonas
  - The Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas